CLINICAL TRIAL: NCT02885506
Title: A Phase I Study to Investigate the Safety, Tolerability and Pharmacokinetic Profile and Food Effect of P218 in Healthy Adult Volunteers
Brief Title: A FIH Study to Investigate the Safety, Tolerability and PK of P218
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMV_P218_15_01; 2016-001933-29 (EudraCT Number)
Record Dates: First submitted 2016-08-19; First posted 2016-08-31 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-05

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Part A of the study was conducted as a dose escalation, and that Part B utilized a cross-over design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Cohort 1 (Experimental): Oral administration of P218 capsules 10 mg
  Interventions: Drug: Oral administration of P218 capsules
- Cohort 2 (Experimental): Oral administration of P218 capsules 30 mg
  Interventions: Drug: Oral administration of P218 capsules
- Cohort 3 (Experimental): Oral administration of P218 capsules 100 mg
  Interventions: Drug: Oral administration of P218 capsules
- Cohort 4 (Experimental): Oral administration of P218 capsules 250 mg
  Interventions: Drug: Oral administration of P218 capsules
- Cohort 5 (Experimental): Oral administration of P218 capsules 500 mg
  Interventions: Drug: Oral administration of P218 capsules
- Cohort 6 (Experimental): Oral administration of P218 capsules 750 mg
  Interventions: Drug: Oral administration of P218 capsules
- Cohort 7 (Experimental): Oral administration of P218 capsules 1000 mg
  Interventions: Drug: Oral administration of P218 capsules
- Cohort 8 - Pooled Placebo (Placebo Comparator): Oral administration of P218 matching placebo
  Interventions: Drug: Oral administration of P218 matching placebo
- Fed - Fasted (Experimental): Oral administration of P218 capsules 250 mg Under fed then fasted conditions.
  Interventions: Drug: Oral administration of P218 capsules
- Fasted - Fed (Experimental): Oral administration of P218 capsules 250 mg Under fasted then fed conditions.
  Interventions: Drug: Oral administration of P218 capsules

INTERVENTIONS:
Drug: Oral administration of P218 capsules — Oral administration of P218 capsules. The number of capsules is determined by the dose level of the cohort.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6; Cohort 7; Fasted - Fed; Fed - Fasted
Drug: Oral administration of P218 matching placebo — Oral administration of P218 matching placebo. The number of capsules is identical to the corresponding number of P218 capsules administered to the volunteers on the investigational drug.
  Arms: Cohort 8 - Pooled Placebo

SUMMARY:
The First in Human (FIH) study is separated into two parts:

* The first part is a Single Ascending Dose (SAD), double-blinded, randomized and placebo-controlled, including 8 cohorts of 8 subjects (2 placebo and 6 on active drug).
* The second part is a food effect cohort with an open-labelled, randomized fed/fasted cross-over design.

The main objectives of the study are to confirm safety, tolerability and Pharmacokinetics (PK) of P218 in healthy volunteers.

DETAILED DESCRIPTION:
The study is divided into two parts:

Part A

This is a double-blind randomised, placebo-controlled, parallel group, ascending dose study and will comprise up to eight fasted cohorts (8 volunteers in each) that will receive a single ascending dose (SAD) of P218 to assess its safety, tolerability and pharmacokinetic profile. Each subject will participate in only one dose group and will receive only one dose of study drug. In each cohort, 2 and 6 subjects will be randomized to placebo and P218, respectively. The data obtained from each cohort will undergo a formal review by the Safety Review Team (SRT). SRT will confirm that it is safe to proceed with the next dose/cohort.

Part B

This is the pilot food effect evaluation. Once predicted human efficacious concentrations of P218 and a safe exposure window (at least 3-fold above the targeted therapeutic exposure in order to account for a possible increase in exposure with food) has been achieved in Part A, a new cohort of 8 subjects (all receiving active drug) will be evaluated for food effect in an open-label, randomized fed/fasted crossover design. Subjects participating in this food effect cohort will be randomized to two single dose sessions (fed/fasted). The second dose will be administered after a washout period of at least 5x observed human half-life (T1/2), to be confirmed once PK data are available from the relevant doses from Part A.

Primary objectives:

* To investigate the safety and tolerability of single escalating oral doses of P218 when administered to healthy volunteers (men and Women of Non Child Bearing Potential (WNCBP)) under fasted conditions.

Secondary objectives:

* To describe the pharmacokinetics of P218 and its major glucuronide metabolite (P218 acyl glucuronide) in healthy volunteers (men and WNCBP) after administration of single escalating oral doses
* To investigate the effect of a high fat meal on the pharmacokinetics and safety/tolerability of P218.

This study incorporates the use of an adaptive design. All anticipated dosing levels can be adjusted in accordance with PK, safety and tolerability data collected up to the decision making time-point.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a healthy male or female (of non-childbearing potential), aged 18 to 45 years, inclusive.
2. Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead electrocardiograms (ECG), and clinical laboratory evaluation (haematology, biochemistry, coagulation, and urinalysis) that is reasonably likely to interfere with the subject's participation in or ability to complete the study as assessed by the Investigator.
3. Subject has a body weight of at least 50 kg and a Body Mass Index (BMI) of 18-25 Kg/m2, inclusive.
4. Female subjects must be of non-childbearing potential:

   1. Natural (spontaneous) post-menopausal defined as being amenorrheic for at least 12 months without an alternative medical cause with a screening follicle stimulating hormone level > 25 IU/L (or at the local laboratory levels for post-menopause).
   2. Premenopausal with irreversible surgical sterilization by hysterectomy and/or bilateral oophorectomy or salpingectomy at least 6 months before screening (as determined by subject medical history).
5. Heterosexually active male subjects with a female spouse/partner of childbearing potential must agree to use barrier contraception (male condom), even with documented medical assessment of surgical success of a vasectomy, if your partner could become pregnant from the time of the first administration of P218 and for 100 days following this. Your partner must also use a method of highly effective contraception including:

   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

     * Oral
     * Intravaginal
     * Transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation:

     * Oral
     * Injectable
     * Implantable
   * Intrauterine device
   * Intrauterine hormone-releasing system
   * Bilateral tubal occlusion
6. Subjects are non-smokers or ex-smokers for more than 90 days prior to screening or smoke no more than 5 cigarettes per day. If users of nicotine products (i.e. spray, patch, e-cigarette, etc.) no more than 5 cigarettes per day is allowed. Subjects must agree to abstain from smoking while in the unit.
7. Ability to swallow multiple capsules at a time or (consecutively) 1 capsule at a time.
8. Subjects must be capable of fully understanding and complying with the requirements of the study and must have signed the informed consent form prior to undergoing any study-related procedures.
9. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Male subjects with a female partner(s) who is (are) pregnant or lactating from the time of the administration of study medication.
2. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means.
3. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal (including gallbladder), cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug or food allergies, anaphylaxis or other severe allergic reactions but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
4. Current or relevant history of physical or psychiatric illness that may require treatment or make the subject unlikely to fully comply with the requirements or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
5. Any surgical or medical condition possibly affecting drug absorption (e.g. cholecystectomy, gastrectomy, bowel disease, etc.), distribution, metabolism or excretion.
6. Any history of gallbladder disease, including cholecystitis and/or cholelithiasis.
7. Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of the participation in the study may influence the result of the study, or the subject's ability to participate in the study.
8. History of photosensitivity.
9. History of megaloblastic anaemia or folate deficiency.
10. History or clinical evidence of substance and/or alcohol abuse within the 12 months before screening. Alcohol abuse is defined as regular weekly intake of more than 21 units for males and 14 units for females (using alcohol tracker http://www.nhs.uk/Tools/Pages/NHSAlcoholtracker.aspx).
11. Treatment with an investigational drug within 90 days or 5 half-lives preceding the first dose of study medication (or as determined by the local requirement, whichever is the longer).
12. Donation of blood or blood products (excluding plasma) within 90 days prior to study medication administration.
13. Use of moderate/strong inhibitors or inducers of Cytochromes P450 (CYP450) or transporters within 30 days or 5 half-lives (whichever is the longer) prior to the first dose of study medication.
14. Consumption of grapefruit, grapefruit juice or grapefruit-related citrus fruits (e.g. Seville oranges, pomelos) within 30 days prior to the first dose of study medication.
15. Ingestion of any poppy seeds within the 24 hours prior to screening.
16. Use of prescription or non-prescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is the longer) prior to the first dose of study medication. With the exception of paracetamol, which may be used incidentally or for a short-term treatment at a maximum dose of 1 gr. per day.
17. Use of herbal supplements at least 30 days prior to the first dose of study medication.
18. Any clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations conducted at screening or on admission.
19. The history or presence of any of the following cardiac conditions: known structural cardiac abnormalities; family history of long QT syndrome; cardiac syncope or recurrent, idiopathic syncope; exercise related clinically significant cardiac events.

    * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of corrected QT interval (QTc) changes. This includes subjects with any of the following (at screening):
    * Sinus node dysfunction.
    * Clinically significant interval prolongation of the interval from the beginning of the P wave to the beginning of the three distinct waves created by the passage of the cardiac electrical impulse through the ventricles (QRS complex) on an electrocardiogram (PR).
    * Intermittent second or third degree atrioventricular (AV) block.
    * Incomplete or complete bundle branch block.
    * Abnormal T wave morphology.
    * Prolonged QT intervals calculated using Bazett's formula (QTcB) >450 ms or shortened QTcB < 350 ms. Any other ECG abnormalities in the standard 12-lead ECG and 24-hour 12 lead Holter ECG or an equivalent assessment which in the opinion of the Investigator will interfere with the ECG analysis.

    Subjects with borderline abnormalities may be included if the deviations do not pose a safety risk, and if agreed between the appointed Cardiologist and the PI.
20. Confirmed positive results from urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates, and methadone) or from the alcohol breath test at screening or on admission.
21. A positive human immunodeficiency virus (HIV) I and II antibodies, hepatitis B surface antigen (HBsAg), anti Hepatitis core antibody (anti hepatitis B core antigen (HBc) immunoglobulin G (IgG) [and anti HBc Immunoglobulin M (IgM) if IgG is positive]), or hepatitis C virus (HCV) antibody at screening.
22. Subjects have veins unsuitable for intravenous puncture or cannulation on either arm (e.g. veins that are difficult to locate access or puncture veins with a tendency to rupture during or after puncture).
23. Any conditions which in the opinion of the investigator would make the subject unsuitable for enrollment or could interfere with the subjects' participation in or completion of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rossignol, PhD, Study Director — Medicines for Malaria Venture
Locations (1):
- Richmond Pharmacology Ltd, Croydon, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 10 mg P218 oral administration
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
- Cohort 2: 30 mg P218 oral administration
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
- Cohort 3: 100 mg P218 oral administration
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
- Cohort 4: 250 mg P218 oral administration
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
- Cohort 5: 500 mg P218 oral administration
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
- Cohort 6: 750 mg P218 oral administration
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
- Cohort 7: 1000 mg P218 oral administration
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
- Pooled Placebo: Placebo capsule oral administration
  Oral administration of P218 matching placebo: The number of capsules is identical to the corresponding number of P218 capsules administered to the volunteers on the investigational drug.
- Fed - Fasted: 250 mg P218 oral administration under fed then fasted conditions.
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
- Fasted - Fed: 250 mg P218 oral administration under fasted then fed conditions.
Period: Part A
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fed - Fasted | Fasted - Fed
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fed - Fasted | Fasted - Fed
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fed - Fasted: A single oral dose of 250 mg of P218 under fed then fasted conditions.
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
- Fasted - Fed: A single oral dose of 250 mg of P218 under fasted then fed conditions.
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fed - Fasted | Fasted - Fed | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 4 | 4 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The study contained two parts, and separate participants were included in each part.
  years
    Part A: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 0 | 0 | 56
    Part A | 32.2 (8.8) | 26.8 (6.9) | 29.7 (8) | 27.2 (7.7) | 26.2 (6.2) | 27.5 (4.1) | 28.7 (7.6) | 25.4 (6.2) |  |  | 27.6 (6.8)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 8
    Part B |  |  |  |  |  |  |  |  | 23 (5) | 32 (6.2) | 27.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The study contained two parts, and separate participants were included in each part.
  Participants
    Part A: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 0 | 0 | 56
    Part A: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0
    Part A: Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 |  |  | 56
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 8
    Part B: Female |  |  |  |  |  |  |  |  | 0 | 0 | 0
    Part B: Male |  |  |  |  |  |  |  |  | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The study contained two parts, and separate participants were included in each part.
  Participants
    Part A: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 0 | 0 | 56
    Part A: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0
    Part A: Asian | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 |  |  | 6
    Part A: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0
    Part A: Black or African American | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 3 |  |  | 8
    Part A: White | 5 | 3 | 4 | 3 | 3 | 5 | 5 | 8 |  |  | 36
    Part A: More than one race | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 |  |  | 6
    Part A: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 8
    Part B: American Indian or Alaska Native |  |  |  |  |  |  |  |  | 0 | 0 | 0
    Part B: Asian |  |  |  |  |  |  |  |  | 0 | 0 | 0
    Part B: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  |  | 0 | 0 | 0
    Part B: Black or African American |  |  |  |  |  |  |  |  | 1 | 1 | 2
    Part B: White |  |  |  |  |  |  |  |  | 3 | 3 | 6
    Part B: More than one race |  |  |  |  |  |  |  |  | 0 | 0 | 0
    Part B: Unknown or Not Reported |  |  |  |  |  |  |  |  | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Population: The study contained two parts, and separate participants were included in each part.
  kg/m²
    Part A: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 0 | 0 | 56
    Part A | 23.2 (1.44) | 22.48 (2) | 23 (1.89) | 23.15 (2.04) | 23 (2.43) | 22.35 (1.74) | 22.57 (2.36) | 21.91 (1.87) |  |  | 22.59 (1.91)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 8
    Part B |  |  |  |  |  |  |  |  | 21.65 (2.52) | 24.65 (1.29) | 23.15 (2.45)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of P218: Incidence, Severity and Relationship to the Investigational Product of Observed and Self-reported Adverse Events
Description: Number of participants with adverse events
Time Frame: During 11 days post administration of a single oral dose of P218 to healthy volunteers
Population: In Part A, forty-two subjects received P218 at single doses of 10, 30, 100, 250, 500, 750 or 1000 mg and 14 subjects received placebo (two each per dose level).
  In Part B, four subjects received a single dose of 250 mg when fasted in Period 1 and fed in Period 2, four other subjects received 250 mg when fed in Period 1 and fasted in Period 2.
Measure: Count of Participants; unit: Participants
Groups:
- Fasted Cohort: A single oral dose of 250 mg of P218 under fasted conditions.
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
- Fed Cohort: A single oral dose of 250 mg of P218 under fed conditions.
  Oral administration of P218 capsules: The number of capsules is determined by the dose level of the cohort.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fasted Cohort | Fed Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 8 | 8
Participants | 0 | 0 | 2 | 1 | 2 | 3 | 3 | 3 | 0 | 1

2. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Measurable Concentration (AUClast)
Description: Estimation of the following PK parameter (in fasted and fed cohorts) using non-compartmental methods: AUClast
Time Frame: During 11 days post administration of a single oral dose of P218 to healthy volunteers
Population: Plasma concentration data were available from all completed cohorts for P218. Hence no data was analysed from the Pooled Placebo cohort.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fasted Cohort | Fed Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 8 | 8
ng.h/mL | 129.799 (34.394) | 443.774 (91.790) | 1610.743 (351.794) | 4007.975 (1017.207) | 8101.229 (2905.479) | 13592.017 (2405.709) | 18286.115 (5915.260) |  | 3409.601 (1062.776) | 3397.972 (1377.368)

3. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: Estimation of the following PK parameter (in fasted and fed cohorts) using non-compartmental methods: AUCinf
Time Frame: During 11 days post administration of a single oral dose of P218 to healthy volunteers
Population: Plasma concentration data available from all completed cohorts for P218. Hence no data analysed for Pooled Placebo cohort.
  Subject 202 in cohort 2 (30 mg) reported a half-life estimate of 19.2 hours, considered outlying with regard to the remainder of the cohort with a geometric mean half-life of 3.13 hrs.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fed - Fasted | Fasted - Fed
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 6 | 5 | 6 | 0 | 8 | 8
h*ng/mL | 133.561 (37.598) | 417.496 (62.144) | 1621.068 (390.845) | 4027.181 (1014.917) | 8126.550 (2904.536) | 13782.492 (2614.899) | 18445.724 (5774.322) |  | 3449.478 (1381.293) | 3440.498 (1055.743)

4. Secondary Outcome: Maximum Plasma Drug Concentration (Cmax)
Description: Estimation of the following PK parameter (in fasted and fed cohorts) using non-compartmental methods: Cmax
Time Frame: During 11 days post administration of a single oral dose of P218 to healthy volunteers
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fed - Fasted | Fasted - Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 8 | 8
ng/mL | 72.567 (38.099) | 208.167 (51.573) | 1000.333 (393.963) | 2120.000 (373.310) | 4441.667 (1799.493) | 6251.667 (1894.027) | 9005.000 (3055.943) |  | 1271.000 (814.827) | 1785.625 (924.390)

5. Secondary Outcome: Time to Reach Maximum (Peak) Plasma Concentration Following Drug Administration (Tmax)
Description: Estimation of the following PK parameter (in fasted and fed cohorts) using non-compartmental methods: Tmax
Time Frame: During 11 days post administration of a single oral dose of P218 to healthy volunteers
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fed - Fasted | Fasted - Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 8 | 8
hours | 1.092 (0.490) | 1.167 (0.408) | 0.917 (0.585) | 1.172 (0.684) | 1.419 (0.668) | 1.589 (1.284) | 1.169 (0.407) |  | 2.500 (1.309) | 1.188 (0.530)

6. Secondary Outcome: Elimination Half-life (t1/2)
Description: Estimation of the following PK parameter (in fasted and fed cohorts) using non-compartmental methods: t1/2
Time Frame: During 11 days post administration of a single oral dose of P218 to healthy volunteers
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fed - Fasted | Fasted - Fed
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 6 | 5 | 6 | 0 | 8 | 8
hours | 3.525 (2.238) | 8.538 (6.492) | 17.615 (4.382) | 12.014 (9.829) | 14.359 (7.666) | 18.314 (11.527) | 24.407 (19.509) |  | 26.007 (12.678) | 23.386 (15.689)

7. Secondary Outcome: Apparent Total Clearance of the Drug From Plasma After Oral Administration (CL/F) (for Parent Only)
Description: Estimation of the following PK parameter (in fasted and fed cohorts) using non-compartmental methods: CL/F (for parent only)
Time Frame: During 11 days post administration of a single oral dose of P218 to healthy volunteers
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fed - Fasted | Fasted - Fed
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 6 | 5 | 6 | 0 | 8 | 8
L/h | 79.978 (22.039) | 73.397 (12.995) | 65.323 (19.235) | 65.292 (15.468) | 67.082 (19.245) | 56.220 (12.022) | 57.812 (14.131) |  | 83598.839 (35344.849) | 78876.051 (24043.587)

8. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase After Oral Administration (Vz/F) (for Parent Only).
Description: Estimation of the following PK parameter (in fasted and fed cohorts) using non-compartmental methods: Vz/F (for parent only).
Time Frame: During 11 days post administration of a single oral dose of P218 to healthy volunteers
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fed - Fasted | Fasted - Fed
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 6 | 5 | 6 | 0 | 8 | 8
L | 371.147 (141.081) | 856.018 (563.080) | 1701.469 (860.918) | 1130.341 (976.613) | 1383.792 (1006.067) | 1618.045 (1431.351) | 2141.443 (2200.839) |  | 2960.939 (1263.797) | 2561.542 (1407.629)

ADVERSE EVENTS:
Time Frame: Up to D29 or longer according to half life.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Pooled Placebo | Fasted Cohort | Fed Cohort
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/14 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/14 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 2/6 | 1/6 | 2/6 | 3/6 | 3/6 | 3/14 | 0/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6) | Cohort 3 (N=6) | Cohort 4 (N=6) | Cohort 5 (N=6) | Cohort 6 (N=6) | Cohort 7 (N=6) | Pooled Placebo (N=14) | Fasted Cohort (N=8) | Fed Cohort (N=8)
PRESYNCOPE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FAECES SOFT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Richmond shall not issue or submit any press release for publication without MMV's prior written approval. In recognition that Richmond and the Site Principal Investigator have a responsibility to ensure that results of scientific interest arising from a Clinical Trial are appropriately published and disseminated, Richmond may, upon MMV's written consent which will not be unreasonably withheld, publish Results of a clinical trial carried out under a Project Agreement.

DOCUMENTS (2):
  • Study Protocol (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT02885506/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT02885506/SAP_001.pdf